CLINICAL TRIAL: NCT03871270
Title: The National Institutes of Health Measure of Healing Experience of All Life Stressors (NIH-HEALS): Factor Analysis and Validation
Brief Title: The National Institutes of Health Measure of Healing Experience of All Life Stressors
Acronym: NIH-HEALS
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Ann Berger, M.D., MSN, MD, National Institutes of Health Clinical Center (CC)
Other Study IDs: 17-CC-00125
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Severe Chronic Illness
Keywords: healing; spiritual; psycho-social-spiritual; growth; chronic illness; patient care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Those with severe chronic illnesses, which included but were not limited to various forms of advanced cancer, blood dyscrasias, graft vs. host disease, and rare genetic conditions.

SUMMARY:
NIH-Healing Experience in All Life Stressors (NIH-HEALS) is a 35 item self-report questionnaire developed by the NIH Clinical Center Pain and Palliative care. It assesses an individual's mechanisms for coping as a means to reach "healing" during life's difficult situations and/or life limiting challenges. The factorial structure of the tool has been recently re-examined with 200 patients. The three main factors are: Connection (including religious, spiritual, interpersonal), Reflection/ Introspection, and Trust/Acceptance.

DETAILED DESCRIPTION:
At the Clinical Center Pain and Palliative Care Service (PPCS) we have developed a pscyho-social-spiritual measure, the Healing Experience in all Life Stressors (HEALS), that focuses on the healing experience in people with severe and life limiting illness. We have validated this tool further in order to be able to identify those individuals who may benefit from additional interventions to cope with their illness and even assist them in reaching a healing experience that is possible even in the midst of their unfavorable circumstances. Identification of vulnerable individuals as well individuals who do have transformative experience after being diagnosed with severe and life limiting illness, has far-reaching impact on the quality of patient care for the very sick patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or above
* The ability to read and write in English
* The presence or history of a serious and/or life-threatening disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients had a history of a serious chronic illness and were already involved in experimental treatments and research projects for the study and treatment of their particular disease at the NIH Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health- Healing Experience of All Life Stressors (NIH-HEALS) | 7 months
  Based on our validation study (Ameli et.al., 2018), we now propose a 35-item, three-factor NIH-HEALS as a measure of psycho-social-spiritual healing. These three factors include: Connection, Reflection & Introspection, and Trust & Acceptance.
Self Integration Scale (SIS) -V2 | 7 months
  SIS is an 18 item self report measure with 2 factors: Healed and Co-dependent. As predicted NIH-HEALS positively correlated with the Healed and negative correlated with the Co-dependent factors.
Functional Assessment of Chronic Illness Therapy-Spiritual well being (FACIT-SP) | 7 months
  FACIT-SP is a 12 item self report that measures spiritual well being and is a part of the larger FACIT measurement system (www.FACIT.org). A 3 factor structure has been reported with cancer patients and include meaning, peace, and faith. As predicted, NIH-HEALS correlated positively with these 3 factors.
Mindful Attention Awareness Scale (MAAS) | 7 months
  MAAS is a self report measure of trait mindfulness with 15 items. As predicted NIH-HEALS correlated positively with MAAS.
The Connor-Davidson Resilience Scale (CD-RISC) (10 item version) | 7 months
  CD-RSIC is a 10 item self-report measure of resilience. As predicted NIH-HEALS positively correlated with CD-RISC
Life Events Checklist 5 (LEC-5) (standard self-report) | 7 months
  LEC-5 is a 17 item self-report measure designed to screen for potentially traumatic events in a respondent's lifetime. The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items.
Demographic Questionnaire (DQ) | 7 months
  DQ collected information on gender, age, ethnicity, race, marital status, religious affiliation, education, employment status, medical diagnosis, length of illness, severity of illness, psychiatric co-morbidity, perceived stress level, perceived level of social support, overall health status, and overall quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Egnew TR. The meaning of healing: transcending suffering. Ann Fam Med. 2005 May-Jun;3(3):255-62. doi: 10.1370/afm.313. PMID 15928230
- [Background] Park CL. Making sense of the meaning literature: an integrative review of meaning making and its effects on adjustment to stressful life events. Psychol Bull. 2010 Mar;136(2):257-301. doi: 10.1037/a0018301. PMID 20192563
- [Background] Skeath P, Norris S, Katheria V, White J, Baker K, Handel D, Sternberg E, Pollack J, Groninger H, Phillips J, Berger A. The nature of life-transforming changes among cancer survivors. Qual Health Res. 2013 Sep;23(9):1155-67. doi: 10.1177/1049732313499074. Epub 2013 Jul 17. PMID 23863850
- [Background] Sloan DH, BrintzenhofeSzoc K, Kichline T, Baker K, Pinzon JP, Tafe C, Li L, Cheng MJ, Berger A. An assessment of meaning in life-threatening illness: development of the Healing Experience in All Life Stressors (HEALS). Patient Relat Outcome Meas. 2017 Feb 16;8:15-21. doi: 10.2147/PROM.S118696. eCollection 2017. PMID 28243158
- [Background] Young WC, Nadarajah SR, Berger AM. Supportive medical care in life-threatening illness: A pilot study. Palliat Support Care. 2016 Dec;14(6):680-685. doi: 10.1017/S147895151600033X. Epub 2016 May 24. PMID 27215292
- [Result] Ameli R, Sinaii N, Luna MJ, Cheringal J, Gril B, Berger A. The National Institutes of Health measure of Healing Experience of All Life Stressors (NIH-HEALS): Factor analysis and validation. PLoS One. 2018 Dec 12;13(12):e0207820. doi: 10.1371/journal.pone.0207820. eCollection 2018. PMID 30540764